CLINICAL TRIAL: NCT03129113
Title: A Multicentre, 48 Week Randomised Controlled Factorial Trial of Adding Maraviroc and/or Metformin for Hepatic Steatosis in HIV-1-infected Adults on Combination Antiretroviral Therapy.
Brief Title: Adding MAraViroc &/or METformin for Hepatic Steatosis in People Living With HIV
Acronym: MAVMET
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); ViiV Healthcare (Industry); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, ADAM CURSLEY, Trial Manager, University College, London
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MAVMET
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Hepatic Steatosis; HIV-1-infection
MeSH Terms: conditions — Fatty Liver | interventions — Maraviroc; Metformin

STUDY DESIGN:
Intervention Model Description: 2 by 2 factorial randomisation to one of the 4 arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- maraviroc (Arm A) (Experimental): maraviroc dosed BID p/o (dose adjusted depending on background combination antiretroviral therapy).
  Interventions: Drug: Maraviroc
- metformin (Arm B) (Experimental): metformin 500mg BID p/o.
  Interventions: Drug: Metformin
- maraviroc + metformin (Arm C) (Experimental): maraviroc dosed BID p/o (dose adjusted depending on background combination antiretroviral therapy) PLUS metformin 500mg BID p/o.
  Interventions: Drug: Maraviroc; Drug: Metformin
- no adjunctive therapy (Arm D) (No Intervention): no adjunctive therapy

INTERVENTIONS:
Drug: Maraviroc — 1:1:1:1 randomisation to one of four arms for 48 weeks
  Arms: maraviroc (Arm A); maraviroc + metformin (Arm C)
Drug: Metformin — 1:1:1:1 randomisation to one of four arms for 48 weeks
  Arms: maraviroc + metformin (Arm C); metformin (Arm B)

SUMMARY:
This is a multicentre, phase IV, randomised, open-label, trial exploring adjunctive maraviroc and/or metformin for liver steatosis over 48 weeks.

Sponsored by University College London Coordinated by MRC Clinical Trials Unit at UCL

DETAILED DESCRIPTION:
There is a global epidemic of obesity and/or being overweight. Fatty liver disease associated with overweight/obesity, can cause liver inflammation, which can lead to scarring of the liver (cirrhosis), liver cancer and early death. It is predicted that fatty liver disease will become the number one cause of liver cirrhosis in the next 20 years. There are no effective treatments, except weight loss, which is rarely successful.

In HIV-infected individuals, antiretroviral therapy (ART) is very successful at maintaining health long-term. However, despite this, data suggest that HIV-infected individuals are at greater risk of developing fatty liver disease than the general population, even if they are not overweight. Past exposure to some of the older, now obsolete, ART drugs, may have added to this greater risk. What makes things more difficult is that fatty liver disease can be 'silent' with no symptoms or signs until quite advanced.

MAVMET is trying to find out if maraviroc (licensed anti-HIV drug) and metformin (licensed for diabetes), given separately or in combination will reduce the amount of liver fat.

MAVMET participants are HIV-infected adult (aged at least 35), with HIV (but not hepatitis B/C) for 5 years or more, on combination ART for at least 1 year, and likely - because of abnormal liver tests and/or a large waist to have increased liver fat or already have a confirmed diagnosis of fatty liver disease, on a previous scan or a liver biopsy.

Participants will continue on their current ART and be randomised (like the flip of a coin) to receive 48 weeks of maraviroc (Arm A) or metformin (Arm B) or both drugs (Arm C) or no additional drugs (Arm D). Participants have 7 clinic visits over 48 weeks to monitor progress and 2 magnetic liver scans (MRI) (no radiation) at University College Hospital to measure liver fat. Mortimer Market Centre participants can also have optional brain MRI at the Institute of Neurology.

Patients can enrol at one of 3 sites: Mortimer Market Centre, St.Thomas's Hospital, King's College Hospital, London.

ELIGIBILITY:
PATIENT INCLUSION CRITERIA

1. Signed informed consent
2. Males or females ≥35 years of age
3. Chronic HIV-1-infection for ≥5 years
4. On combination antiretroviral therapy (cART) and with virological suppression (<50 copies/mL) for ≥1 year
5. i) >1 abnormal (above the upper limit) of LFTS (ALT or AST) in the last 2 years with no other explanation (e.g. secondary syphilis) and/or ii) increased waist circumference ≥94 cm (≥90cm if South Asian origin) in men, ≥80cm in women and/or iii) a confirmed diagnosis of NAFLD on liver imaging (CT/MRI/ultrasound), FibroScan and/or iv) liver biopsy confirmed diagnosis of NALFD
6. Females of child bearing potential (CBP) who agree to avoid pregnancy for the duration of the trial
7. Able to comply with protocol requirements

PATIENT EXCLUSION CRITERIA

1. Co-infection with hepatitis B or C
2. Confirmed chronic liver disease from any other cause (e.g. hepatitis C, hepatitis B)
3. Daily intake of alcohol >20g in women and >30g in men
4. Current illicit drug use that in the opinion of the investigator would interfere with patient's ability to comply with the protocol
5. On metformin or another biguanide agent;
6. Currently on maraviroc
7. Any contraindication to the receipt of maraviroc and/or metformin
8. Known B12 deficiency
9. Pregnant or breast feeding
10. Contraindication to MRI scanning
11. Peanut or soya allergy
12. eGFR <60 ml/min/1.73m2
13. ALT ≥10 x ULN
14. History of cardiovascular (ischaemic heart disease) or cerebrovascular disease.
15. Any other condition that in the opinion of the investigator would not make the patient suitable for the trial.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Change in percentage of liver fat as measured by MR PDFF between baseline and week 48. | 48 weeks
  MR PDFF

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pett, Principal Investigator — UCL
Locations (6):
- United Kingdom (6):
  - Royal London Hospital, London
  - Royal Free Hospital, London
  - St Thomas' Hospital, London
  - King's College Hospital, London
  - St Mary's Hospital, London
  - UCL Mortimer Market Centre, London

IPD SHARING:
Plan to Share IPD: No